CLINICAL TRIAL: NCT06929949
Title: A Single-center, Prospective, Observational Cohort Study on the Effect of Different Digestive Tract Reconstruction Methods on Postoperative Quality of Life After Proximal Gastrectomy
Brief Title: The Effect of Different Digestive Tract Reconstruction Methods on Postoperative Quality of Life After Proximal Gastrectomy
Acronym: STARS-GC10
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Director, Clinical Professor, The First Hospital of Jilin University
Other Study IDs: STARS-GC10
Record Dates: First submitted 2025-03-12; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Junction (GEJ) Cancer; Gastric Cancer
Keywords: Robot-assisted surgery; Laparoscopic-assisted surgery; Proximal gastrectomy; Digestive tract reconstruction
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Double-flap technique (DFT): The DFT digestive tract reconstruction was performed in patients with gastric cancer after proximal gastrectomy
- double-tract reconstruction (DTR): The DTR digestive tract reconstruction was performed in patients with gastric cancer after proximal gastrectomy
- Tubular gastric anastomosis (TGA): The TGA digestive tract reconstruction was performed in patients with gastroesophageal cancer after proximal gastrectomy

SUMMARY:
Gastric cancer ranks as the fifth most common malignancy worldwide and the fourth leading cause of cancer-related deaths. In China, its incidence and mortality rank third among all cancers. While the global incidence of gastric cancer is declining, proximal gastric cancer and adenocarcinoma of the esophagogastric junction (AEG) are on the rise. Due to the unique characteristics of AEG, there is no standardized treatment consensus, making the selection of an optimal surgical approach and reconstruction method crucial for improving patient outcomes.

For early-stage proximal gastric cancer and AEG, total gastrectomy (TG) and proximal gastrectomy (PG) are common surgical options. PG, increasingly favored for its function-preserving benefits, has been shown to be a safe and effective alternative to TG. While TG effectively removes lymph nodes and reduces reflux risk, it leads to permanent loss of gastric function and nutritional deficiencies. PG better preserves gastrointestinal function but is limited by the risk of reflux esophagitis, highlighting the need for improved reconstruction techniques.

Several reconstruction methods exist after PG, including esophagogastric anastomosis, jejunal interposition, double-tract reconstruction (DTR), double-flap technique (DFT), and tubular gastric anastomosis, each with varying efficacy in preventing reflux. Studies suggest that DTR reduces reflux and improves quality of life compared to esophagogastric anastomosis, while DFT, first introduced in 1998, has gained popularity for its advantages in maintaining nutrition and minimizing reflux. Additionally, tubular gastric anastomosis, which constructs a narrow gastric tube to facilitate tension-free anastomosis, has shown potential benefits for AEG patients.

Most existing studies on laparoscopic or robot-assisted reconstruction techniques for proximal gastric cancer are retrospective, lacking high-quality prospective evidence. Furthermore, comparative data on their anti-reflux efficacy and postoperative quality of life remains l

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common malignant tumor worldwide and ranks fourth in cancer-related mortality. In China, the incidence and mortality rate of gastric cancer rank third among all malignancies. While the global incidence of gastric cancer has been steadily declining, the incidence of proximal gastric cancer has been rising. Additionally, the incidence of adenocarcinoma of the esophagogastric junction (AEG) has been increasing annually, showing an upward trend worldwide. Due to its unique anatomical location and significant tumor biological heterogeneity, there is no standardized consensus on the optimal treatment for AEG. Therefore, selecting an appropriate surgical resection and reconstruction approach remains crucial for improving the prognosis of patients with proximal gastric cancer and AEG.

For early-stage proximal gastric cancer and AEG, either total gastrectomy (TG) or proximal gastrectomy (PG) can be performed. With the advancement of function-preserving surgical concepts, PG has been increasingly recognized as a viable option. The Japanese Clinical Oncology Group (JCOG1401) trial demonstrated that laparoscopic proximal gastrectomy (LPG) is a safe and effective treatment for early-stage proximal gastric cancer compared to laparoscopic total gastrectomy (LTG). However, patients undergoing TG often experience long-term postoperative quality-of-life concerns. Although TG can effectively remove lymph nodes and reduce the risk of gastroesophageal reflux, it results in the permanent loss of gastric storage, mechanical grinding, and secretory functions, as well as reduced feasibility of postoperative endoscopic examination. TG patients may also suffer from nutritional deficiencies, including vitamin B12 deficiency, iron deficiency, weight loss, anemia, diarrhea, and dumping syndrome. In contrast, PG offers advantages in preserving gastrointestinal function and nutritional status. However, its widespread adoption is limited by the risk of reflux esophagitis. Thus, selecting an optimal reconstruct

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years.
* Preoperative gastroscopic pathological biopsy was performed, and histologically confirmed as carcinoma (papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, poorly differentiated adenocarcinoma, mixed adenocarcinoma, etc.) or adenoma.
* Diagnosed with upper gastric cancer (T1N0M0, T1N1M0, or T2N0M0) or esophagogastric junction cancer with a diameter ≤4 cm based on the 8th edition of the AJCC staging system, as confirmed by CT, MRI, endoscopic ultrasound, and pathology.
* Undergoing proximal gastrectomy with D2 lymphadenectomy is expected to achieve curative resection, with the remaining gastric volume required to be at least half of the pre-resection volume.
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale.
* ASA (American Society of Anesthesiology) class I to III.
* The patient has adequate organ function and is capable of tolerating surgery.
* Written informed consent.

Exclusion Criteria:

* Patients who have received preoperative radiotherapy, chemotherapy, targeted therapy, or immunotherapy.
* Presence of multiple malignant tumors in the stomach.
* History of upper abdominal surgery, except for laparoscopic cholecystectomy.
* History of gastric surgery, except for endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR) for gastric cancer.
* Evidence of distant metastasis diagnosed by thoracoabdominal CT/MRI or PET-CT.
* Pregnant or lactating women.
* History of uncontrolled epilepsy, central nervous system disorders, or psychiatric illness.
* Patients with limb disabilities or motor function impairment.
* History of other malignant diseases within the past five years, except for cured skin cancer and cervical carcinoma in situ.
* Clinically severe (i.e., active) heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or higher congestive heart failure, severe arrhythmia requiring medical intervention, or myocardial infarction within the past six months.
* History of stroke or cerebral hemorrhage within the past six months.
* Severe, uncontrolled recurrent infections or other serious uncontrolled comorbidities.
* Pulmonary function test showing FEV1 < 50% of the predicted value.
* Patients requiring emergency surgery due to tumor-related complications (e.g., bleeding, perforation, or obstruction).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper gastric cancer (T1N0M0, T1N1M0, or T2N0M0 according to the AJCC 8th edition) and esophageal junction cancer (≤4cm in diameter).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2028-11-25 (Estimated); Study Completion 2030-11-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of reflux esophagitis | Follow-up evaluations are performed up to 2 years postoperatively.
  The proportion of patients with reflux esophagitis diagnosed by digestive endoscopy (LA classification), barium meal (barium meal) and (GerdQ scale).

SECONDARY OUTCOMES:
Incidence of Postoperative complications | Within 30 days after surgery
  The total number of patients who underwent surgical treatment was used as the denominator, and the number of patients with any postoperative complication was used as the numerator to calculate the incidence percentage.
Postoperative mortality | Within 30 days after surgery
  The total number of patients who underwent surgical treatment was used as the denominator, and the number of patients who died after surgery was used as the numerator to calculate the incidence percentage.
Body weight change | Follow-up evaluations are performed up to 2 years postoperatively.
  Body weight will be monitored during follow-up after surgery.
Long-term postoperative quality of life | Follow-up evaluations are performed up to 2 years postoperatively.
  Quality of life was assessed by EORTC QLQ-STO22 questionnaires.
Long-term postoperative quality of life | Follow-up evaluations are performed up to 2 years postoperatively.
  Quality of life was assessed by EORTC QLQ-C30 questionnaires.
Postoperative albumin | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Postoperative prealbumin | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Postoperative total protein | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Postoperative hemoglobin | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Vitamin D | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Folic acid | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Vitamin B12 | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Ferritin | Follow-up evaluations are performed up to 2 years postoperatively.
  Hematological examination
Sarcopenia | Follow-up evaluations are performed up to 2 years postoperatively.
  CT scan was performed to assess the L3 skeletal muscle index (LSMI).
Hp Infection | Follow-up evaluations are performed up to 2 years postoperatively.
  C13/14 examination by blowing or by endoscopic biopsy.
3-years Relapse free survival rate | Follow-up evaluations are performed up to 3 years postoperatively.
3-years overall survival rate | Follow-up evaluations are performed up to 3 years postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Muraoka A, Kobayashi M, Kokudo Y. Laparoscopy-Assisted Proximal Gastrectomy with the Hinged Double Flap Method. World J Surg. 2016 Oct;40(10):2419-24. doi: 10.1007/s00268-016-3510-5. PMID 27094564
- [Background] Kuroda S, Nishizaki M, Kikuchi S, Noma K, Tanabe S, Kagawa S, Shirakawa Y, Fujiwara T. Double-Flap Technique as an Antireflux Procedure in Esophagogastrostomy after Proximal Gastrectomy. J Am Coll Surg. 2016 Aug;223(2):e7-e13. doi: 10.1016/j.jamcollsurg.2016.04.041. Epub 2016 May 6. No abstract available. PMID 27157920
- [Background] Zhang Y, Zhang H, Yan Y, Ji K, Jia Z, Yang H, Fan B, Wang A, Wu X, Zhang J, Ji J, Ji X, Bu Z. Double-tract reconstruction is superior to esophagogastrostomy in controlling reflux esophagitis and enhancing quality of life after proximal gastrectomy: Results from a prospective randomized controlled clinical trial in China. Chin J Cancer Res. 2023 Dec 30;35(6):645-659. doi: 10.21147/j.issn.1000-9604.2023.06.09. PMID 38204447
- [Background] Park DJ, Han SU, Hyung WJ, Hwang SH, Hur H, Yang HK, Lee HJ, Kim HI, Kong SH, Kim YW, Lee HH, Kim BS, Park YK, Lee YJ, Ahn SH, Lee I, Suh YS, Park JH, Ahn S, Park YS, Kim HH. Effect of Laparoscopic Proximal Gastrectomy With Double-Tract Reconstruction vs Total Gastrectomy on Hemoglobin Level and Vitamin B12 Supplementation in Upper-Third Early Gastric Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2256004. doi: 10.1001/jamanetworkopen.2022.56004. PMID 36790808
- [Background] Cho M, Son T, Kim HI, Noh SH, Choi S, Seo WJ, Roh CK, Hyung WJ. Similar hematologic and nutritional outcomes after proximal gastrectomy with double-tract reconstruction in comparison to total gastrectomy for early upper gastric cancer. Surg Endosc. 2019 Jun;33(6):1757-1768. doi: 10.1007/s00464-018-6448-x. Epub 2018 Sep 10. PMID 30203207
- [Background] Jung DH, Lee Y, Kim DW, Park YS, Ahn SH, Park DJ, Kim HH. Laparoscopic proximal gastrectomy with double tract reconstruction is superior to laparoscopic total gastrectomy for proximal early gastric cancer. Surg Endosc. 2017 Oct;31(10):3961-3969. doi: 10.1007/s00464-017-5429-9. Epub 2017 Mar 24. PMID 28342130
- [Background] Katai H, Mizusawa J, Katayama H, Kunisaki C, Sakuramoto S, Inaki N, Kinoshita T, Iwasaki Y, Misawa K, Takiguchi N, Kaji M, Okitsu H, Yoshikawa T, Terashima M; Stomach Cancer Study Group of Japan Clinical Oncology Group. Single-arm confirmatory trial of laparoscopy-assisted total or proximal gastrectomy with nodal dissection for clinical stage I gastric cancer: Japan Clinical Oncology Group study JCOG1401. Gastric Cancer. 2019 Sep;22(5):999-1008. doi: 10.1007/s10120-019-00929-9. Epub 2019 Feb 20. PMID 30788750
- [Background] Yamasaki M, Takiguchi S, Omori T, Hirao M, Imamura H, Fujitani K, Tamura S, Akamaru Y, Kishi K, Fujita J, Hirao T, Demura K, Matsuyama J, Takeno A, Ebisui C, Takachi K, Takayama O, Fukunaga H, Okada K, Adachi S, Fukuda S, Matsuura N, Saito T, Takahashi T, Kurokawa Y, Yano M, Eguchi H, Doki Y. Multicenter prospective trial of total gastrectomy versus proximal gastrectomy for upper third cT1 gastric cancer. Gastric Cancer. 2021 Mar;24(2):535-543. doi: 10.1007/s10120-020-01129-6. Epub 2020 Oct 29. PMID 33118118